CLINICAL TRIAL: NCT03482323
Title: Improving Survival in Lung Cancer Patients: A Randomized Controlled Trial of Aerobic Exercise and Tai-chi Interventions
Brief Title: Aerobic Exercise and Tai-chi Interventions for Improving Survival in Lung Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Chia-Chin Lin, Head of School of Nursing, Alice Ho Miu Ling Nethersole Charity Foundation Professor in Nursing, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UW18154
Record Dates: First submitted 2018-03-22; First posted 2018-03-29 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Lung Cancer Patients
MeSH Terms: interventions — Exercise; Tai Ji

STUDY DESIGN:
Intervention Model Description: The participants will be randomised into equally sized arms; tai-chi classes, exercise classes, or control.
Who Masked: Outcomes Assessor
Masking Description: All baseline and follow-up assessments will be carried out by research staff who are blinded to allocation. The statistician and laboratory staff for the measurement of biomarkers remains still blinded until the end of the whole study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise intervention (Experimental): Exercise class will run twice a week for 12 weeks. Participants will be encouraged to maintain their exercise beyond the intervention. An exercise trainer will lead the classes. The main activity of the classes includes aerobic exercises of walking on treadmill, or out-doors depending on group preference and weather, at a set pace individually tailored for moderate intensity of exercise, determined by baseline physical functioning assessment and modified based on Rated Perceived Exertion (RPE), or cycling on a stationary bike, using a set resistance to the physical functioning assessment and RPE. A set of four strengthening exercises are included in one of the exercise classes each week. These exercises are chosen to increase strength in the leg, arm, abdomen and improve trunk stability. Weights for the strengthening exercise will be set to give participants a moderate level of intensity of exercise.
  Interventions: Behavioral: Exercise
- Tai-chi intervention (Experimental): The classes will run twice a week for 12 weeks with each session lasting approximately 60 minutes. Classes will be taught by an experienced tai-chi master, who will explain the theory behind tai-chi and the principles of the techniques. The supervised session includes a warm up, self-massage and a guided run through of the movements, breathing techniques, and relaxation in tai-chi. The tai-chi master will guide participants to practice the tai-chi they learn in the classes at home each day. Upon completion of the 12 weeks course, participants will be encouraged to continue their tai-chi practice, given guidance on local services and programmes they may join if they wish to.
  Interventions: Behavioral: Tai-Chi
- Control group (No Intervention): Participants randomised to the control group shall receive written information on health levels of physical activity, which they can participate in at home (self-management) and continue to receive their usual care, participants will be followed up with an assessment at 12 weeks, 6 months and one year. At the end of the evaluation stage of the study, survivors in the control group will be invited to take part in an intervention of their choice.

INTERVENTIONS:
Behavioral: Exercise — Our exercise class intervention is based on current best evidence and will be tailored for each participant's ability for exercise. The exercise classes is also designed to fit into the guidelines for exercise in adults aged 18 years and above with a long term health condition. During the 12 weeks in the training, exercises will be varied (mixing up time spent on bikes and walking) along with the intensities of exercise varied to keep the classes more engaging for participants and maintaining compliance to the programme.
  Arms: Exercise intervention
Behavioral: Tai-Chi — Our tai-chi classes will be based on a 24-form Yang style of tai-chi exercise set.
  Arms: Tai-chi intervention

SUMMARY:
This proposed study aims to examine the effect of classical aerobic exercise or tai-chi on 1-year survival rate of lung cancer patients compared to usual care, as a primary outcome of this study. To understand the hypothesized outcomes of improved survival of lung cancer patients through physical exercise or tai-chi practice intervention, we will examine the changes in some subjective psychosocial outcomes and objective biomarkers that may be associated with the survival of cancer patients, as the secondary outcome of this study. Those biomarkers will be in following aspects: 1.) circadian rhythm, 2.) cardio-respiratory fitness, and 3.) immune functions. Secondary outcome measures include: quality of life, psychological distress, quality of sleep, fatigue, level of physical activity, circadian rhythms, cardio-respiratory fitness, physical functioning tests and immune function. The pilot study aims to assess the feasibility and acceptability of the trial so that the main study will have a higher chance of success.

DETAILED DESCRIPTION:
Lung cancer is one of the commonest cancers around the world. The current prognosis for lung cancer is poor, with a 1-year survival rate of only 42%. Thus, lung cancer imposes a substantial health burden on patients and society both locally and world widely. On top of the classical clinical therapies, additional approaches that could result in survival benefit are needed.

Previous studies, including our own, have shown that physical exercise, such as aerobic walking, improves lung cancer patient's physical fitness particularly cardiovascular fitness, circadian rhythm and immune function. Another popular mode of exercise in Chinese population is tai-chi. With emphasis on breathing and concentration, tai-chi exhibits extra benefits for stress-relieving and psychological well-being. Those benefits of exercise have long been implicated for better survival of cancer patients. The promising benefits of aerobic exercise or tai-chi, as non-pharmacological interventions, urge for need of rigorous evidence on the effectiveness of these interventions in improving survival outcomes. However, to date, there has been no report from a randomized controlled trial (RCT) to study the effect of aerobic exercise or tai-chi on survival of lung cancer patients.

This proposed research is designed to conduct a three-arm RCT comparing aerobic exercise, tai-chi to usual care in non-small cell lung cancer patients. Recruited participants will be randomised into three groups: 1) a 12-week aerobic exercise group, 2) a 12-week tai-chi program group, and 3) a self-management control group. Aerobic exercise and tai-chi program will be conducted by certificated coaches. Life-long adherence to the practice in intervention groups is encouraged.

Through this project we aim to evaluate if 1) aerobic exercise or 2) tai-chi intervention increases survival (measured by 1-year survival rate) in lung cancer patients compared to control, as the primary outcome of this study. We shall also examine if tai-chi practice can provide similar survival benefits compared with ordinary exercise. Using biomarkers including circadian rhythm, cardio-respiratory fitness, and immune function further provides objective measures for bio-physiological effectiveness of the interventions. The associations of those biological measures and psycho-social status with survival outcomes will be further explored.

Findings of this study will provide crucial information on the evidence-based practice by physical exercise or tai-chi to improve survival of lung cancer patients. This study will also have far-reaching significance in providing important scientific evidence to policymakers to integrate physical activity into routine clinical management as an add-on treatment for lung cancer patients in Hong Kong.

The pilot study aims to assess the feasibility and acceptability (such as attendance, drop out, satisfaction) of the trial so that the main study will have a higher chance of success.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are diagnosed of stage IIIB, or IV non-small-cell lung cancer confirmed by pathology
2. Patients are not currently engaged in other research or participant in any other exercise or mind-body classes
3. Patients aged 18 years old, or above
4. Patients who can communicate in Cantonese, Mandarin or English
5. Patients with no other cancer diagnosis within the previous 1 year
6. Patients report not doing regular exercises (defined <150 min of moderate-intensity exercise weekly) in daily living, but are able to attend either exercise or tai-chi classes at scheduled times
7. Patients being conscious and alert.

Exclusion Criteria:

Patients suffering from a diagnosed active neurological, substance abuse and /or psychiatric disorders (i.e. depression, chronic insomnia) will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
One-year survival rate | One year
  Duration of survival in participants shall be monitored. For cases of death, causes of death will be collected from patients' clinical dataset to insure data quality. Cancer progress-free survival will be taken at the end of the study period.

SECONDARY OUTCOMES:
Levels of physical activity | Baseline, 12 weeks, 6 months and one year
  To measure compliance to exercise all participants will be measured for their level of physical activity in daily living. Physical activity will be quantified with a non-invasive small-size wrist-worn piezoelectric accelerometer (Actigraph; Ambulatory Monitoring Inc., New York). Actigraphy has been shown to provide valid assessments of physical activity. The user-defined time interval for the count of wrist accelerations is 1 min. Patients will be asked to wear the actigraph for at least 3 consecutive 24-hour spans. Each patient will keep a diary for times of rising and retiring.
Circadian rhythms- cortisol and melatonin rhythms | Baseline and one year
  We will measure circadian rhythms using biomarkers that have been linked to survival of cancer patients, melatonin rhythms and cortisol rhythms will be measured using saliva samples collected before and after intervention. The melatonin and cortisol levels will be measured using enzyme-linked immunosorbent assay (ELISA) kits. The saliva will be collected using Salivettes at following time points: 1 hour, 6 hour, 12 hour and 16 hour after habitual wake time (referred as circadian time).
Cardio-respiratory fitness- 6-minute walking test | Baseline, 12 weeks, 6 months and one year
  Cardio-respiratory fitness shall be evaluated using the 6-minute walking test (6MWT). The 6MWT has been widely used to assess cardio-respiratory fitness in lung cancer patients [28-30]. The 6MWT requires participants to walk on an even and flat surface between two cones set 30m apart, with the object being the participant walking as far as possible within the 6 minutes period (if participant cannot continue for the 6 minutes, the test will end). The walking test is measured in units of meters walked at the end of the 6 minutes.
Physical functioning- timed up and go test, sit to stand test, single leg standing test, Get Active Questionnaire | Baseline, 12 weeks, 6 months and one year
  A battery of physical functioning tests will be used to evaluate participants' agility (timed up and go test), strength (sit to stand test) and balance (single leg standing test). Physical fitness will also be assessed using the Get Active Questionnaire (GAQ). The GAQ assesses if participants are safe to participate in the interventions and ensures if participants can perform the exercises within the intervention.
Immune functions- cytotoxic activity of natural killer (NK) cells, and spontaneous or phytohemagglutinin (PHA)-stimulated T-lymphocyte proliferation | Baseline and one year
  For each participant, 10 ml of peripheral blood will be collected before and after intervention in intervention groups, as well as in control group at the same time points, for some immune functional studies. The peripheral blood mononuclear cells are isolated for measurements of immune functions. Immune functions will be analyzed by cytotoxic activity of natural killer (NK) cells, and spontaneous or phytohemagglutinin (PHA)-stimulated T-lymphocyte proliferation
Health-related quality of Life- European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire and the corresponding lung cancer-specific module | Baseline, 12 weeks, 6 months and one year
  Health related QoL is an important outcome for lung cancer patients and plays an important impact on prognosis. The Chinese version of the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30) and the corresponding lung cancer-specific module (QLQ-LC13) shall be used as measurements of QoL
Psychological Distress- Hospital Anxiety and Depression Score | Baseline, 12 weeks, 6 months and one year
  To evaluate psychological distress the Hospital Anxiety and Depression Score (HADS) will be used. The HADS comprises seven items each for anxiety and depression. Each item of the anxiety subscale and the depression subscale was scored on a 4-point scale. This scale is a reliable tool, and is widely used to assess patients with cancer.
Quality of Sleep (Subjective)- Pittsburgh Sleep Quality Index | Baseline, 12 weeks, 6 months and one year
  To assess quality of sleep, the Chinese version of the Pittsburgh Sleep Quality Index (PSQI) shall be used. This instrument has been used worldwide to assess patients' perceived sleep quality in both clinical and research. The results have supported the psychometric properties of the PSQI.
Fatigue- Brief Fatigue Inventory | Baseline, 12 weeks, 6 months and one year
  Fatigue will be measured by the Chinese version of the Brief Fatigue Inventory (BFI). The BFI was developed to measure fatigue in cancer patients. It consists of 9 items with each item scored on a 0-10 scale. The BFI measures patients' fatigue when symptoms are at their worst, least, usual and currently during the normal waking hours, with 0 indicating no fatigue, and 10 being fatigue as bad as one can imagine. Other items include fatigues interaction with patients' general activity, mood, waking ability, normal work (includes both work outside the home and housework), relations with other people, ability to think clearly, and enjoyment of life. The interference is measured with 0 being does not interfere, and 10 being completely interferes.
Quality of Sleep (Objective)- Actigraph | Baseline, 12 weeks, 6 months and one year
  Actigraph will serve as an objective measure for assessing sleep parameters, such as sleep efficiency, total sleep time.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Chin Lin, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Background] Fong DY, Ho JW, Hui BP, Lee AM, Macfarlane DJ, Leung SS, Cerin E, Chan WY, Leung IP, Lam SH, Taylor AJ, Cheng KK. Physical activity for cancer survivors: meta-analysis of randomised controlled trials. BMJ. 2012 Jan 30;344:e70. doi: 10.1136/bmj.e70. PMID 22294757
- [Background] Mustian KM, Katula JA, Gill DL, Roscoe JA, Lang D, Murphy K. Tai Chi Chuan, health-related quality of life and self-esteem: a randomized trial with breast cancer survivors. Support Care Cancer. 2004 Dec;12(12):871-6. doi: 10.1007/s00520-004-0682-6. Epub 2004 Sep 30. PMID 15599776
- [Background] Sui X, Lee DC, Matthews CE, Adams SA, Hebert JR, Church TS, Lee CD, Blair SN. Influence of cardiorespiratory fitness on lung cancer mortality. Med Sci Sports Exerc. 2010 May;42(5):872-8. doi: 10.1249/MSS.0b013e3181c47b65. PMID 19996990
- [Background] Chen HM, Tsai CM, Wu YC, Lin KC, Lin CC. Effect of walking on circadian rhythms and sleep quality of patients with lung cancer: a randomised controlled trial. Br J Cancer. 2016 Nov 22;115(11):1304-1312. doi: 10.1038/bjc.2016.356. Epub 2016 Nov 3. PMID 27811855
- [Background] Chen HM, Tsai CM, Wu YC, Lin KC, Lin CC. Randomised controlled trial on the effectiveness of home-based walking exercise on anxiety, depression and cancer-related symptoms in patients with lung cancer. Br J Cancer. 2015 Feb 3;112(3):438-45. doi: 10.1038/bjc.2014.612. Epub 2014 Dec 9. PMID 25490525
- [Derived] Cheung DST, Takemura N, Lam TC, Ho JCM, Deng W, Smith R, Yan Y, Lee AWM, Lin CC. Feasibility of Aerobic Exercise and Tai-Chi Interventions in Advanced Lung Cancer Patients: A Randomized Controlled Trial. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211033352. doi: 10.1177/15347354211033352. PMID 34549648
- [Derived] Takemura N, Cheung DST, Fong DYT, Lee AWM, Lam TC, Ho JC, Kam TY, Chik JYK, Lin CC. Relationship of subjective and objective sleep measures with physical performance in advanced-stage lung cancer patients. Sci Rep. 2021 Aug 26;11(1):17208. doi: 10.1038/s41598-021-96481-7. PMID 34446756